CLINICAL TRIAL: NCT04125680
Title: Community-Based Participatory English as a Second Language Health Literacy Program to Prevent Lead Exposure in Flint
Brief Title: English as a Second Language Health Literacy Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: ACE Community Health (Other); Genesee County Hispanic Latino Collaborative (Other); National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Emily Feuerherm, Associate Professor, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HUM #00148555; UL1TR002240 (NIH)
Record Dates: First submitted 2019-10-03; First posted 2019-10-14 (Actual); Results first posted 2023-02-24 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Health Literacy; Language
MeSH Terms: conditions — Language

STUDY DESIGN:
Intervention Model Description: A pilot trial will be used: study participants will be registered and placed into the program on a first-come, first-served basis. This will result in a study assessing correlation rather than causation.
Masking Description: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ESL Health Literacy Classes (Other): The program will last 8 weeks with classes held online during evening hours. The curriculum will focus on using pedagogies for health literacy as a practice. Assessments will be administered pre-post intervention.
  Interventions: Behavioral: ESL Health Literacy Classes

INTERVENTIONS:
Behavioral: ESL Health Literacy Classes — The intervention will last 8-weeks, and the first and last classes will be devoted to survey assessments. Participants will be asked to reflect on their health knowledge and behaviors, and how they have changed since starting the program. The curriculum administered during the classes will use pedagogies for health literacy as a practice. It will focus on skills needed to learn about lead exposure in the ESL classroom: (1) vocabulary; (2) grammar; and (3) identifying risk factors, symptoms and preventive strategies. A focus on health literacy as practice will include personal engagement using language in context: (1) role-play interactions about lead exposure prevention; (2) discussing views about risk, and how to talk about it with peers and family members; (3) identifying sources of reliable health information; and (4) learning to ask for support and resources.

SUMMARY:
This research is using a Community-Based Participatory Action Research (CBPAR) approach to design, implement, and evaluate English as a Second Language health literacy classes for Hispanic adults to reduce lead exposure.

DETAILED DESCRIPTION:
This Community-Based Participatory Action Research (CBPAR) aims to:

1. Develop a community-based participatory English as a Second Language (ESL) health literacy curriculum for lead exposure that can be used in other locations or programs.
2. Determine the outcomes of the curriculum, including changes in knowledge about lead, access to health resources, and health behavioral changes to reduce lead exposure.
3. To evaluate the implementation of the ESL health literacy curriculum.

This research focuses on ESL health literacy classes provided to Hispanic adults to reduce lead exposure. This research will use a pilot test with a pre-post test design. The program will last for 8 weeks; with weeks 1 and 8 as the assessment weeks. The curriculum uses pedagogies that move participants from health literacy as functional skill to health literacy as social practice where knowledge is used for empowerment and meaningful change. The goals of this research are to demonstrate increased health literacy knowledge, improved health behaviors, increased access to health services, and improved English language proficiency for Hispanic residents of Flint in relation to lead exposure prevention.

ELIGIBILITY:
Inclusion Criteria:

* Hispanic immigrants living in or around Flint.
* Native speakers of Spanish, with varying degrees of English fluency and literacy.
* 18 years old and older.

Exclusion Criteria:

* Immigrants from other linguistic backgrounds will be excluded at this time because all program materials will be bilingually available in English and Spanish.
* Children will be excluded at this time because we are focusing on ESL health literacy for adults.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2021-05-20 (Actual); Primary Completion 2021-09-15 (Actual); Study Completion 2021-09-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emily Feuerherm, PhD, Principal Investigator — University of Michigan-Flint
Locations (1):
- University of Michigan - Flint, Flint, Michigan, United States

REFERENCES:
- [Derived] Baumeister A, Aldin A, Chakraverty D, Hubner C, Adams A, Monsef I, Skoetz N, Kalbe E, Woopen C. Interventions for improving health literacy in migrants. Cochrane Database Syst Rev. 2023 Nov 14;11(11):CD013303. doi: 10.1002/14651858.CD013303.pub2. PMID 37963101

RESULTS

PARTICIPANT FLOW:
Groups:
- ESL Health Literacy Classes: The program will last 5-8 weeks with classes held online during evening hours. The curriculum will focus on using pedagogies for health literacy as a practice. Assessments will be administered pre-post intervention.
  ESL Health Literacy Classes: The intervention will last 5-8 weeks, and the first and last classes will be devoted to survey assessments. Participants will be asked to reflect on their health knowledge and behaviors, and how they have changed since starting the program. The curriculum administered during the classes will use pedagogies for health literacy as a practice. It will focus on skills needed to learn about lead exposure in the ESL classroom: (1) vocabulary; (2) grammar; and (3) identifying risk factors, symptoms and preventive strategies. A focus on health literacy as practice will include personal engagement using language in context: (1) role-play interactions about lead exposure prevention; (2) discussing views about risk, and how to talk about it with peers and family members; (3) identifying sources of reliable health information; and (4) learning to ask for support and resources.
Period: Overall Study
Arm/Group | ESL Health Literacy Classes
Started | 17
Completed | 2
Not Completed | 15
Not completed — Lost to Follow-up | 15

BASELINE CHARACTERISTICS:
Arm/Group | ESL Health Literacy Classes
Number analyzed (Participants) | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.21 (9.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Practicing Safe Lead Exposure Prevention Behaviors (Pre Test)
Description: ESL Hispanic adult learners' lead exposure prevention adherence to the evidence-based recommendations set by the Environmental Protection Agency (EPA) and the Centre for Disease Control and Prevention (CDC) for reducing exposure to water containing levels of lead above 15 ppb for the use was measured using a 3 item questionnaire. Questions include: (1) I have had my water tested for lead; (2) I have an NSF approved filter for my drinking water; and (3) I use bottled water or water from a filtration system for drinking and cooking to reduce or eliminate my lead exposure. Response options are yes, no and don't know. The numbers below represent participants who answered 'Yes' to each question.
Time Frame: Baseline
Population: Five people participated in the health literacy curriculum which is where this outcome was measured.
Measure: Count of Participants; unit: Participants
Groups:
- ESL Health Literacy Classes: The program will last up to 8 weeks with classes held online during evening hours. The curriculum will focus on using pedagogies for health literacy as a practice. Assessments will be administered pre-post intervention.
  ESL Health Literacy Classes: The intervention will last up to 8 weeks, and the first and last classes will be devoted to survey assessments. Participants will be asked to reflect on their health knowledge and behaviors, and how they have changed since starting the program. The curriculum administered during the classes will use pedagogies for health literacy as a practice. It will focus on skills needed to learn about lead exposure in the ESL classroom: (1) vocabulary; (2) grammar; and (3) identifying risk factors, symptoms and preventive strategies. A focus on health literacy as practice will include personal engagement using language in context: (1) role-play interactions about lead exposure prevention; (2) discussing views about risk, and how to talk about it with peers and family members; (3) identifying sources of reliable health information; and (4) learning to ask for support and resources.
Arm/Group | ESL Health Literacy Classes
Number analyzed (Participants) | 5
Participants
  I have had my water tested for lead. | 1
  I have an NSF-approved filter for my drinking water. | 2
  I use bottled water or water from a filtration system to reduce or eliminate my lead exposure | 5

2. Primary Outcome: Number of Participants Practicing Safe Lead Exposure Prevention Behaviors (Post Test)
Description: as for outcome 1
Time Frame: Up to 8-weeks post-treatment
Population: Five people participated in the health literacy curriculum which is where this outcome was measured.
Measure: Count of Participants; unit: Participants
Arm/Group | ESL Health Literacy Classes
Number analyzed (Participants) | 5
Participants
  I have had my water tested for lead. | 3
  I have an NSF-approved filter for my drinking water. | 5
  I use bottled water or water from a filtration system to reduce or eliminate my lead exposure | 5

3. Secondary Outcome: Lead Exposure Prevention Knowledge (Pre-Test)
Description: ESL Hispanic adult learners' lead exposure prevention knowledge of the evidence-based recommendations set by the EPA and the CDC for reducing exposure to water containing levels of lead above 15 ppb. Numerical score measured by questions on the Chicago Lead Knowledge Test questionnaire. Five questions related to the 24 question Chicago Lead Knowledge test questionnaire were administered to participants. One point was assigned to each correct response. A participant could earn five total points; with five total points meaning all questions were answered correctly. A composite value was created for the 5 questions.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ESL Health Literacy Classes
Number analyzed (Participants) | 17
units on a scale | 3.35 (0.86)

4. Secondary Outcome: Lead Exposure Prevention Knowledge (Post Test)
Description: as for outcome 3
Time Frame: Up to 8-weeks post-treatment
Population: Only two participants were administered and completed the post test. Due to the COVID-19 pandemic overall enrollment in the study was low and several participants withdrew from the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ESL Health Literacy Classes
Number analyzed (Participants) | 2
units on a scale | 4 (0)

5. Secondary Outcome: Health Literacy Level (Pre-Test)
Description: ESL Hispanic adult learner's health literacy score. Numerical score measured by questions on the Fostering Literacy for Good Health Today (FLIGHT) Nive Desarollando Amplia Salud (VIDAS) Test.
  The short 10-question FLIGHT VIDAS test was administered to participants in Spanish. One point was assigned to each correct response. A participant could earn 10 total points. The literacy level scale is: 0-3 below basic, 4-6 basic, 7-8 intermediate, 9-10 proficient.
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | ESL Health Literacy Classes
Number analyzed (Participants) | 17
Participants
  Below basic literacy (0-3 correct answers) | 3
  Basic literacy (4-6 correct answers) | 5
  Intermediate literacy (7-8 correct answers) | 3
  Proficient literacy (9-10 correct answers) | 6

6. Secondary Outcome: Health Literacy Level (Post-Test)
Description: ESL Hispanic adult learner's health literacy score. Numerical score measured by questions on the Fostering Literacy for Good Health Today (FLIGHT) Nive Desarollando Amplia Salud (VIDAS) Test.
Time Frame: Up to 8-weeks post-treatment
Population: Responses to the post test literacy questions not available because the FLIGHT/VIDAS was a separate test and the post test was not administered due to study team oversight.
Arm/Group | ESL Health Literacy Classes
Number analyzed (Participants) | 0

7. Other Pre Specified Outcome: Number of Participants Who Experienced Food Insecurity as Measured by the National Health and Nutrition Examination Survey (Pre Test)
Description: ESL Hispanic adult learners' level of food security was measured using two questions from the National Health and Nutrition Examination Survey. The questions include: (1) In the past 12 months how often did you or anyone else in your household worry there would not be enough to eat because of a lack of money and (2) In the past 12 months how often did you or anyone else in your household not eat quality or variety of foods that you wanted to eat because of a lack of money. Possible response options include 'Often', 'Sometimes', 'Never', 'Don't Know', and 'Refuse to Answer'.
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | ESL Health Literacy Classes
Number analyzed (Participants) | 17
Participants
  How often did you worry that there would not be enough to eat because of a lack of money?: Often | 0
  How often did you worry that there would not be enough to eat because of a lack of money?: Sometimes | 9
  How often did you worry that there would not be enough to eat because of a lack of money?: Never | 4
  How often did you worry that there would not be enough to eat because of a lack of money?: Don't Know | 0
  How often did you worry that there would not be enough to eat because of a lack of money?: Refuse | 4
  How often did you not eat the quality or variety of foods because of a lack of money?: Often | 0
  How often did you not eat the quality or variety of foods because of a lack of money?: Sometimes | 4
  How often did you not eat the quality or variety of foods because of a lack of money?: Never | 9
  How often did you not eat the quality or variety of foods because of a lack of money?: Don't Know | 0
  How often did you not eat the quality or variety of foods because of a lack of money?: Refuse | 4

8. Other Pre Specified Outcome: Number of Participants Who Experienced Food Insecurity as Measured by the National Health and Nutrition Examination Survey (Post Test)
Description: as for outcome 7
Time Frame: Up to 8 weeks post treatment
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | ESL Health Literacy Classes
Number analyzed (Participants) | 2
Participants
  How often did you worry that there would not be enough to eat because of a lack of money?: Often | 0
  How often did you worry that there would not be enough to eat because of a lack of money?: Sometimes | 0
  How often did you worry that there would not be enough to eat because of a lack of money?: Never | 2
  How often did you worry that there would not be enough to eat because of a lack of money?: Don't Know | 0
  How often did you worry that there would not be enough to eat because of a lack of money?: Refuse | 0
  How often did you not eat the quality or variety of foods because of a lack of money?: Often | 0
  How often did you not eat the quality or variety of foods because of a lack of money?: Sometimes | 0
  How often did you not eat the quality or variety of foods because of a lack of money?: Never | 2
  How often did you not eat the quality or variety of foods because of a lack of money?: Don't Know | 0
  How often did you not eat the quality or variety of foods because of a lack of money?: Refuse | 0

9. Other Pre Specified Outcome: Number of Participants Able to Obtain Health Information as Measured by the National Health and Nutrition Examination Survey (Pre Test)
Description: ESL Hispanic adult learners' completed three questions to evaluate their ability to obtain health information. Three questions taken from the National Health and Nutrition Examination Survey were administered to participants. Questions include (1) In the past 12 months did you do anything to improve your health (2) In the past 12 months have you required health information or advice for yourself or a family member and (3) In the past 12 months did you ever experience any difficulties getting the health information or advice for yourself or a family member. Response options are yes, no and don't know. The numbers below represent participants who answered 'Yes' to each question.
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | ESL Health Literacy Classes
Number analyzed (Participants) | 17
Participants
  Did you do anything to improve your health? | 9
  Have you required health information or advice for yourself or a family member? | 8
  Did you ever experience any difficulties getting the health information or advice | 5

10. Other Pre Specified Outcome: Number of Participants Able to Obtain Health Information as Measured by the National Health and Nutrition Examination Survey (Post Test)
Description: as for outcome 9
Time Frame: Up to 8-weeks post-treatment
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | ESL Health Literacy Classes
Number analyzed (Participants) | 2
Participants
  Did you do anything to improve your health? | 0
  Have you required health information or advice for yourself or a family member? | 0
  Did you ever experience any difficulties getting the health information or advice | 0

11. Other Pre Specified Outcome: Perception of Community Belonging as Measured by the National Health and Nutrition Examination Survey (Pre Test)
Description: ESL Hispanic adult learners' were asked to describe their sense of belonging to thier local community. Participants were asked to complete a question taken from the National Health and Nutrition Examination Survey asking them to rate their sense of belonging to their local community from 'very strong' (1) to 'very weak' (4). Responses could include 'very strong','somewhat strong', 'somewhat weak', 'very weak', 'don't know', and 'refuse to answer'. The numbers below represent the participants who selected each response.
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | ESL Health Literacy Classes
Number analyzed (Participants) | 17
Participants
  Very Strong | 0
  Somewhat Strong | 2
  Somewhat Weak | 1
  Very Weak | 10
  Don't Know | 1
  Refused to Answer | 3

12. Other Pre Specified Outcome: Perception of Community Belonging as Measured by the National Health and Nutrition Examination Survey (Post Test)
Description: as for outcome 11
Time Frame: Up to 8 weeks post treatment
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | ESL Health Literacy Classes
Number analyzed (Participants) | 2
Participants
  Very Stong | 0
  Somewhat Strong | 0
  Somewhat Weak | 1
  Very Weak | 0
  Don't Know | 0
  Refused to Answer | 1

13. Other Pre Specified Outcome: Number of Participants With Health Care Coverage as Measured by the Behavioral Risk Factor Surveillance Survey (Pre Test)
Description: ESL Hispanic adult learners' were asked to describe their health care coverage status. Numerical score measured by questions on the Behavioral Risk Factor Surveillance Survey. Participants were asked (1) Do you have any kind of health case coverage including health insurance, prepaid plans such as HMOs, or government plans such as Medicare, or Indian Health Service? Responses could include 'Yes', 'No' and 'Don't Know'. The participants who answered 'Yes' are represented below.
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | ESL Health Literacy Classes
Number analyzed (Participants) | 17
Participants | 7

14. Other Pre Specified Outcome: Number of Participants With Health Care Coverage as Measured by the Behavioral Risk Factor Surveillance Survey (Post Test)
Description: as for outcome 13
Time Frame: Up to 8 weeks post-treatment
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | ESL Health Literacy Classes
Number analyzed (Participants) | 2
Participants | 2

ADVERSE EVENTS:
Time Frame: Up to 8 weeks
Groups:
- ESL Health Literacy Classes: The program will last 5-8 weeks with classes held online during evening hours. The curriculum will focus on using pedagogies for health literacy as a practice. Assessments will be administered pre-post intervention.
  ESL Health Literacy Classes: The intervention will last 5-8-weeks, and the first and last classes will be devoted to survey assessments. Participants will be asked to reflect on their health knowledge and behaviors, and how they have changed since starting the program. The curriculum administered during the classes will use pedagogies for health literacy as a practice. It will focus on skills needed to learn about lead exposure in the ESL classroom: (1) vocabulary; (2) grammar; and (3) identifying risk factors, symptoms and preventive strategies. A focus on health literacy as practice will include personal engagement using language in context: (1) role-play interactions about lead exposure prevention; (2) discussing views about risk, and how to talk about it with peers and family members; (3) identifying sources of reliable health information; and (4) learning to ask for support and resources.
Arm/Group | ESL Health Literacy Classes
All-Cause Mortality (participants affected / at risk) | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17
Other Adverse Events (participants affected / at risk) | 0/17

LIMITATIONS AND CAVEATS:
The main limitation to this study was low enrollment: (1) it was moved online for the pandemic and they preferred in-person, (2) they did not have time or technology to join the online program, and/or (3) interest had waned because of pandemic-related delays, or community-internal politics made some people distrust the community partner.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-04-22): https://cdn.clinicaltrials.gov/large-docs/80/NCT04125680/Prot_SAP_000.pdf
  • Informed Consent Form (2022-04-29): https://cdn.clinicaltrials.gov/large-docs/80/NCT04125680/ICF_001.pdf